CLINICAL TRIAL: NCT03446677
Title: Somatosensory Deficiencies Affect Postural Stability in Asymptomatic Individuals With HIV
Brief Title: Postural Stability Deficiencies in Asymptomatic Individuals With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Martin Rosario, Assistant Professor, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: A2540114
Record Dates: First submitted 2018-02-11; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: HIV; Balance; Vestibular Disorder; Somatosensory Disorders; Postural Stability
Keywords: HIV; Balance; Vestibular; Somatosensory; postural stability; center of pressure
MeSH Terms: conditions — Vestibular Diseases; Somatosensory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asymptomatic persons with HIV (Experimental)
  Interventions: Other: Postural Stability Testing

INTERVENTIONS:
Other: Postural Stability Testing — Each subject was instructed to stand in a static bipedal posture on the MatScan® pressure mat and performed 8 balance tasks. Data of center of pressure, antero-posterior sways and medial-lateral sways were collected in each of the conditions. Each task took 30 seconds to be performed. The first 4 tasks were performed with the mat on the hard surface of the floor. These 4 tasks are as follows: standing with eyes open, standing with eyes closed, standing with eyes open looking and actively moving head upward and downward, and standing with eyes closed and the head actively moving upward and downward. The subjects were asked to perform four more tasks while standing on a thick piece of balance foam that was placed on top of the MatScan®. The remaining 4 tasks are as follows: standing with eyes open, standing with eyes closed, standing with eyes open looking and actively moving the head upward and downward, and standing with eyes closed with head actively moving upward and downward.

SUMMARY:
Persons with HIV can present vestibular system impairments, affecting postural stability. There is scarce literature related to the contribution of the visual and somatosensory systems in maintaining postural stability in persons with HIV. The purpose of this study is to describe the sensory systems used to maintain postural stability and how the sources of sensory information contributes to postural stability in asymptomatic persons with HIV. Postural stability was measured in 20 asymptomatic persons with HIV (11 male, 9 female, aged 43 ± 8 years). Static postural stability was evaluated during eight conditions that perturbed the visual, somatosensory and vestibular inputs. A paired-samples t-test was conducted to compare center of pressure (COP), antero-posterior displacement (APD) and right-left displacement (RLD) on stable and unstable surface and to characterize each balance sensory system. There was a significant difference in the COP and APD of eyes open condition compared to the remaining conditions on stable surface. Furthermore, there was a significant difference in the COP, APD and RLD for the eyes open on a foam surface compared to the remaining conditions on an unstable surface. Postural instability can be detected in asymptomatic persons with HIV under challenging conditions, previous to the evident appearance of balance impairments.

DETAILED DESCRIPTION:
The institutional review boards (IRB) of the University of Puerto Rico Medical Science Campus, reviewed and approved this study before any data collection was initiated. An informed consent was provided to each subject to access their medical records, HIV status, CD4+ cell count and as a requirement to participate in the study.

The subjects were recruited from La Perla de Gran Precio (Community wellness center that specializes in individuals with HIV) localized in San Juan, Puerto Rico. Each subject was evaluated by interview and review of their medical record for the inclusion and exclusion criteria assessment. Different tests were performed as a screening tool to identify additional limitations or impairments in the different sensory systems. To rule out severe neuropathy, the subject had to be able to detect a Semmes- Weinstein Monofilament of 5.07 or less in more than two areas of the foot.12,13 The visual system was screened using Snellen chart and the subject had to obtain at least 20/40 of visual acuity. To rule out severe balance impairments, the Romberg Test and Fukuda's Stepping Test were used. For Romberg Test, subjects had to maintain standing position for 30 seconds and Fukuda's Stepping Test required that the subject did not rotate more than 30° from the initial position or deviate more than 0.5 meters from the center of the circle. Functional strength of lower extremities was screened using a Five Times Sit to Stand test, where the subject had to complete the test in 10 seconds or less. Severe proprioception impairments were assessed using a Proprioceptive Awareness test, where the subject was asked to replicate the initial position performed by the evaluator in the contralateral ankle joint in three trials. After the screening of the inclusion and exclusion criteria, a total of 20 subjects were able to participate in the study.

Each subject was instructed to stand in a static bipedal posture on the MatScan® pressure mat and performed eight balance tasks. Data of center of pressure, antero-posterior sways and medial-lateral sways were collected in each of the conditions. Each task took 30 seconds to be performed. The first four tasks were performed with the mat on the hard surface of the floor. These four tasks are as follows:1) eyes open looking at a fixed point to evaluate all systems (EO); 2) eyes closed (with head fixed approximately 90˚) to eliminate visual input (EC); 3) eyes open looking at a fixed point and actively moving head upward and downward to alter vestibular inputs (EO+HUD). The subject was instructed to maintain a movement frequency of 60bpm and amplitude of approximately 45 degrees in each direction: neck flexion and extension; 4) eyes closed (with head fixed approximately 90˚) to eliminate visual input and the head actively moves upward and downward to alter vestibular inputs (EC+HUD). The subject is instructed to maintain the movement frequency and amplitude as described in task 3.

The subjects were asked to perform four more tasks while standing on a thick piece of balance foam that was placed on top of the MatScan®, creating an unstable surface. The remaining four tasks (tasks 5-8) are as follows: 5) eyes open looking at a fixed point while standing on the balance foam to alter somatosensory inputs (EO+BF); 6) eyes closed with head fixed approximately 90˚ while standing on the balance foam to alter somatosensory inputs and eliminate visual inputs (EC+BF); 7) eyes open looking at a fixed point and actively moving the head upward and downward while standing on the balance foam to alter somatosensory and vestibular inputs (EO+HUD+BF). The subject was instructed to maintain the movement frequency and amplitude as described in task 3; 8) eyes closed with head fixed approximately 90˚ and actively move head upward and downward while standing on the balance foam to eliminate visual inputs and alter somatosensory and vestibular inputs (EC+HUD+BF). The subject is instructed to maintain the movement frequency and amplitude as described in task 3.

Data of postural stability was obtained using the MatScan® pressure mat (TekScan, Boston, MA). The data collected from the pressure mat was analyzed with Tekscan Sway Analysis Module™ (SAM) software (TekScan, Boston, MA) designed for this purpose. Mean and standard deviation were used to describe data. The statistical software used was SPSS-20 to perform a Paired-Samples t-test and compare the center of pressure, antero-posterior and right-left body sways displacement. P values <0.05 were accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. CD4 levels above 300,
2. age within the range of 25-57 years
3. walks without assistive device
4. tolerates standing position for at least 30 minutes
5. stable cardiorespiratory system.

Exclusion Criteria:

1. diagnosis of AIDS (CD4 levels less than 200)
2. diagnosis of Diabetes, Dementia or Arthritis
3. severe neuropathy
4. severe balance impairments
5. severe visual acuity problems that are not treated
6. BMI > 40,
7. decreased functional strength in the lower extremities
8. severe proprioception impairments
9. falls during the last 6 months
10. back or lower extremities lesion or surgery during the last 6 months
11. the use of medications that causes drowsiness 24 hours previous to intervention
12. women that are pregnant or think they might be pregnant

Ages: 25 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07-22 (Actual); Primary Completion 2015-05-22 (Actual); Study Completion 2015-07-22 (Actual)

PRIMARY OUTCOMES:
Postural Stability | Baseline
  Postural stability was operationally defined by the center of pressure displacement measured by the MatScan® pressure mat. These sensors detect the displacement as the body sways anterior, posterior or laterally (right or left).

CONTACTS AND LOCATIONS:
Overall Officials: Martin G Rosario, Ph.D, Principal Investigator — Texas Woman's University

REFERENCES:
- [Background] Sullivan EV, Rosenbloom MJ, Rohlfing T, Kemper CA, Deresinski S, Pfefferbaum A. Pontocerebellar contribution to postural instability and psychomotor slowing in HIV infection without dementia. Brain Imaging Behav. 2011 Mar;5(1):12-24. doi: 10.1007/s11682-010-9107-y. PMID 20872291
- [Background] Heinze BM, Vinck BM, Hofmeyr LM, Swanepoel de W. Vestibular involvement in adults with HIV/AIDS. Auris Nasus Larynx. 2014 Apr;41(2):160-8. doi: 10.1016/j.anl.2013.08.003. Epub 2013 Oct 19. PMID 24145102
- [Background] Cohen HS, Cox C, Springer G, Hoffman HJ, Young MA, Margolick JB, Plankey MW. Prevalence of abnormalities in vestibular function and balance among HIV-seropositive and HIV-seronegative women and men. PLoS One. 2012;7(5):e38419. doi: 10.1371/journal.pone.0038419. Epub 2012 May 31. PMID 22675462
- [Background] Heinze B, Swanepoel DW, Hofmeyr LM. Systematic review of vestibular disorders related to human immunodeficiency virus and acquired immunodeficiency syndrome. J Laryngol Otol. 2011 Sep;125(9):881-90. doi: 10.1017/S0022215111001423. Epub 2011 Jul 5. PMID 21729430
- [Background] Shumway-Cook A, Woollacott M. (2012). Normal Postural Control. In: Motor Control Translating Research into Clinical Practice. 4th ed. Baltimore, MD: Lippincott Williams & Wilkins;:
- [Background] Ruhe A, Fejer R, Walker B. The test-retest reliability of centre of pressure measures in bipedal static task conditions--a systematic review of the literature. Gait Posture. 2010 Oct;32(4):436-45. doi: 10.1016/j.gaitpost.2010.09.012. Epub 2010 Oct 13. PMID 20947353
- [Background] Dellepiane M, Medicina MC, Mora R, Salami A. Static and dynamic posturography in patients with asymptomatic HIV-1 infection and AIDS. Acta Otorhinolaryngol Ital. 2005 Dec;25(6):353-8. PMID 16749603
- [Background] Teggi R, Giordano L, Pistorio V, Bussi M. Vestibular function in HIV patients: preliminary report. Acta Otorhinolaryngol Ital. 2006 Jun;26(3):140-6. PMID 17063983
- [Background] Rosario M, Ortiz A. Balance assessment in people with HIV. Paper presented at: 60th Annual Meeting of American College of Sports Medicine (ACSM)
- [Background] Adamo DE, Pociask FD, Goldberg A. The contribution of head position, standing surface and vision to postural control in young adults. J Vestib Res. 2013;23(1):33-40. doi: 10.3233/VES-130473. PMID 23549053
- [Background] Duffy JC, Patout CA Jr. Management of the insensitive foot in diabetes: lessons learned from Hansen's disease. Mil Med. 1990 Dec;155(12):575-9. PMID 2125335
- [Background] Bell-Krotoski J, Weinstein S, Weinstein C. Testing sensibility, including touch-pressure, two-point discrimination, point localization, and vibration. J Hand Ther. 1993 Apr-Jun;6(2):114-23. doi: 10.1016/s0894-1130(12)80292-4. PMID 8393725
- [Background] FUKUDA T. The stepping test: two phases of the labyrinthine reflex. Acta Otolaryngol. 1959 Mar-Apr;50(2):95-108. doi: 10.3109/00016485909129172. No abstract available. PMID 13636842
- [Background] Whitney SL, Wrisley DM, Marchetti GF, Gee MA, Redfern MS, Furman JM. Clinical measurement of sit-to-stand performance in people with balance disorders: validity of data for the Five-Times-Sit-to-Stand Test. Phys Ther. 2005 Oct;85(10):1034-45. PMID 16180952
- [Background] Chui K, Schmitz T. (2007). Examination of sensory function. In: O'Sullivan S, Schmitz T. Physical Rehabilitation.
- [Background] Heinze BM, Vinck BM, Swanepoel DW. Does the human immunodeficiency virus influence the vestibulocollic reflex pathways? A comparative study. J Laryngol Otol. 2014 Sep;128(9):772-9. doi: 10.1017/S0022215114001996. Epub 2014 Aug 28. PMID 25166876
- [Background] O'Sullivan SB. (2007). Examination of Motor Function: Motor Control and Motor Learning. In: O'Sullivan SB. Physical Rehabilitation. 5th ed. Philadelphia
- [Background] Creath R, Kiemel T, Horak F, Peterka R, Jeka J. A unified view of quiet and perturbed stance: simultaneous co-existing excitable modes. Neurosci Lett. 2005 Mar 29;377(2):75-80. doi: 10.1016/j.neulet.2004.11.071. Epub 2004 Dec 19. PMID 15740840
- [Background] Trenkwalder C, Straube A, Paulus W, Krafczyk S, Schielke E, Einhaupl KM. Postural imbalance: an early sign in HIV-1 infected patients. Eur Arch Psychiatry Clin Neurosci. 1992;241(5):267-72. doi: 10.1007/BF02195975. PMID 1606190
- [Background] Sarlegna FR, Malfait N, Bringoux L, Bourdin C, Vercher JL. Force-field adaptation without proprioception: can vision be used to model limb dynamics? Neuropsychologia. 2010 Jan;48(1):60-7. doi: 10.1016/j.neuropsychologia.2009.08.011. PMID 19695273
- [Background] Cameron M, Monroe L. (2007). Balance and fall risk. In: Tyner T, Allen D. Physical Rehabilitation Evidence-Based Examination, Evaluation, and Intervention. San Louis, Missouri: Saunders. 300-332
- See also: National Institute of health. (2014). Visual acuity test. — http://www.nlm.nih.gov/medlineplus/spanish/ency/article/003396.htm
- See also: Vestibular disorders association. (2009). Vision Challenges with Vestibular Disorders. — http://vestibular.org/sites/default/files/page_files/Vision%20Challenges.pdf